CLINICAL TRIAL: NCT06701760
Title: Exogenous Sodium Lactate Infusion in Traumatic Brain Injury (ELI-TBI)
Brief Title: Sodium Lactate in Severe TBI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Paul Vespa, MD, Professor and Assistant Dean, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20-011590
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; coma; intensive care; brain metabolism
MeSH Terms: conditions — Brain Injuries, Traumatic; Coma | interventions — Sodium Lactate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant is not awake and is not told which arm they were randomized to Assessor is blinded to randomization allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- intervention (Active Comparator): sodium lactate
  Interventions: Drug: Sodium Lactate
- placebo (Placebo Comparator): sodium cbloride infusion
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Sodium Lactate — sodium lactate
  Arms: intervention
Drug: placebo — infusion of sodium chloride
  Other Names: sodium chloride
  Arms: placebo

SUMMARY:
This is a safety phase 2 clinical trial of intravenous infusion of sodium lactate in patients with severe TBI. This study is intended for patients in the acute setting in an intensive care unit at centers that have been selected to participate in this trial. This is a proof of safety study and biomarker response study.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) consists of a primary localized insult to the brain followed by prolonged global disruption of brain metabolism, thus creating risk for secondary brain damage from energy deficiency. To date, there is no specific metabolic treatment to improve outcome after TBI. This study is designed to determine if providing a unique chemical fuel in the form sodium lactate will improve the brain's metabolism and prevent ongoing damage. The investigators will seek to find the highest dose of sodium lactate that is tolerated and then to determine if administering this dose for 24 hours improves brain metabolism and survival. We will collect blood and brain MRI images to test if the intervention helps brain metabolism and brain structure. The study will be a randomized trial so that we have a comparison group against which to best evaluate safety. Ten medical centers that are very experienced with traumatic brain injury will participate in the study and will be supervised by a data safety monitoring board. This is a pilot study that will ultimately inform the design of a large scale clinical trial of sodium lactate in the near future.

RATIONALE TBI has no definitive drug treatment, and multiple trials have failed. We propose a pilot safety study of a metabolic treatment for TBI using exogenous sodium lactate (ELI) infusion to enhance brain oxidative metabolism as a medical treatment for TBI.

STUDY DESIGN This is a multicenter phase 2 study. The phase 2a study will identify the maximum tolerated dose of ELI using the continual reassessment dose escalation design with three dose tiers and will be followed by a phase 2b, randomized, placebo-controlled comparison of the ELI at maximum tolerated dose (MTD) for 24 hours vs normal saline infusion. The time to enrollment and start of study infusion will be 24 hours after onset of TBI.

PRIMARY OBJECTIVE The primary objective of part 1, the dose finding study is to determine the maximum tolerated dose (MTD) associated with a prespecified probability of dose limiting toxicity (DLT). The DLT is defined as the occurrence within 7 days of ELI of any one of three adverse events: AKI, arrythmia (atrial or ventricular tachycardia that causes hypotension), or ARDS (mild or greater).

The primary objective of the part 2 of the study, the randomized trial of MTD ELI for 24 hours vs saline is 30 day mortality.

NUMBER OF SUBJECTS 264

SUBJECT SELECTION

CRITERIA Inclusion Criteria:

1. GCS at enrollment 3-18;
2. Male or female aged 18-80 at admission;
3. acute positive CT findings;
4. ability for subject to comply with the requirements of the study;
5. written informed consent obtained from subject or subject's legal representative.

Exclusion Criteria:

1. Penetrating TBI,
2. Polytrauma leading to instability of systemic hemodynamics, acidosis, or severe acute lung injury during the inclusion period.
3. History of neurological disease, including Parkinson's, Huntington's, Alzheimer's, etc.; History of diabetes mellitus;
4. Serum sodium ≥ 148 mM; Metabolic acidosis pH <7.34;
5. Coagulopathy INR > 1.3, platelets < 100,000, or hematocrit < 28 mg/dl;
6. Renal insufficiency with GFR < 60% of expected or Cr > 1.3;

6. AST or ALT > 1.5x upper limit of normal; Severe liver trauma; 7. baseline serum lactate > 2 mM; 8. Hypotension SBP < 90 refractory to vasopressors; 9. Known mitochondrial genetic disorder; 10. Pregnancy; 11.Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data; 12.Member of a protected population; simultaneous participation in another randomized trial

Time Window Enrollment and study infusion starts within 24 hours of TBI

TEST PRODUCT, DOSE, AND ROUTE OF ADMINISTRATION Sodium Lactate Injection, USP diluted to 200 mg/mL Sodium Lactate.

Lactate will be administered continuously for up to 6 hours by IV (in part 1) and for 24 hours (in part 2) and titrated to achieve targeted blood lactate concentrations for the assigned dose tier. New IND is pending. Investigational Product to be made by Altasciences.

CONTROL PRODUCT, DOSE AND ROUTE OF ADMINISTRATION 0.9% Normal Saline will serve as placebo in part 2 of the study Saline infusion will be administered continuously for up to 24 hours in 24 hours in part 2 of the study

ELIGIBILITY:
Inclusion Criteria:

* GCS at enrollment 3-8
* Male or female aged 18-80 at admission
* acute positive CT findings
* ability for subject to comply with the requirements of the study
* written informed consent obtained from subject or subject's legal representative.

Exclusion Criteria:

* Penetrating TBI
* Polytrauma leading to instability of systemic: hemodynamics, acidosis, or severe acute lung injury during the inclusion period
* History of neurological disease, including Parkinson's, Huntington's, Alzheimer's, etc.
* History of diabetes mellitus
* Serum sodium ≥ 148 mM
* Metabolic acidosis pH <7.34
* Coagulopathy INR > 1.3, platelets < 100,000, or hematocrit < 28 mg/dl
* Renal insufficiency with GFR < 60% of expected or Cr > 1.3;
* AST or ALT > 1.5x upper limit of normal; Severe liver trauma;
* baseline serum lactate > 2 mM
* Hypotension SBP < 90 refractory to vasopressors
* Known mitochondrial genetic disorder
* Pregnancy
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Member of a protected population; simultaneous participation in another randomized trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2028-01-10 (Estimated); Primary Completion 2035-12-30 (Estimated); Study Completion 2038-07-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 30 days
  Mortality
Dose limiting toxicity | 7 days
  panel of serious adverse events

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bernini A, Miroz JP, Abed-Maillard S, Favre E, Iaquaniello C, Ben-Hamouda N, Oddo M. Hypertonic lactate for the treatment of intracranial hypertension in patients with acute brain injury. Sci Rep. 2022 Feb 22;12(1):3035. doi: 10.1038/s41598-022-07129-z. PMID 35194150
- [Result] Wolahan SM, Mao HC, Real C, Vespa PM, Glenn TC. Lactate supplementation in severe traumatic brain injured adults by primed constant infusion of sodium L-lactate. J Neurosci Res. 2018 Apr;96(4):688-695. doi: 10.1002/jnr.24085. Epub 2017 May 20. PMID 28543565
- [Result] Glenn TC, Martin NA, Horning MA, McArthur DL, Hovda DA, Vespa P, Brooks GA. Lactate: brain fuel in human traumatic brain injury: a comparison with normal healthy control subjects. J Neurotrauma. 2015 Jun 1;32(11):820-32. doi: 10.1089/neu.2014.3483. Epub 2015 Mar 31. PMID 25594628
- [Result] Glenn TC, Kelly DF, Boscardin WJ, McArthur DL, Vespa P, Oertel M, Hovda DA, Bergsneider M, Hillered L, Martin NA. Energy dysfunction as a predictor of outcome after moderate or severe head injury: indices of oxygen, glucose, and lactate metabolism. J Cereb Blood Flow Metab. 2003 Oct;23(10):1239-50. doi: 10.1097/01.WCB.0000089833.23606.7F. PMID 14526234